CLINICAL TRIAL: NCT06244160
Title: High Flow Oxygen Therapy After Spinal Cord Injury - Feasibility Study to Design a Pragmatic Randomised Controlled Trial Protocol
Brief Title: High Flow Oxygen Therapy After Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiff and Vale University Health Board (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 8713
Record Dates: First submitted 2023-12-08; First posted 2024-02-06 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Spinal Cord Injuries; Respiratory Failure
MeSH Terms: conditions — Spinal Cord Injuries; Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Feasibility randomised control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): High flow oxygen therapy delivered via nasal cannalue
  Interventions: Other: High flow oxygen therapy
- Control (No Intervention): Standard care with oxygen therapy as required.

INTERVENTIONS:
Other: High flow oxygen therapy — High flow oxygen therapy delivered via nasal cannulae, at 50 litres flow with variable oxygen levels
  Arms: Intervention

SUMMARY:
The goal of this feasibility study is to learn about the ability to use a different form of oxygen therapy (known as high flow oxygen therapy) in patients who have a spinal cord injury in the upper back or neck.

The main questions it aims to answer are:

1. Is it possible to recruit patients to the study
2. It is possible to follow the protocol in its current format
3. What is the impact on those receiving the intervention.

Participants will be randomised to receive either standard care or high flow oxygen therapy for 10 days following inclusion.

DETAILED DESCRIPTION:
In the UK, the annual incidence of acute spinal cord injury (SCI) is 19 new cases per million population, contributing to an estimated 50,000 people who are currently living with SCI1. Trauma is the most common cause of SCI, predominantly from falls and road traffic accidents. Damage to the spinal cord occurs both at the time of injury (primary) and in its aftermath (secondary). Effectively treating and preventing secondary cord injury, and managing complications associated with SCI, can make a significant improvement to patient outcomes.

Respiratory dysfunction is one of the most common medical complications, as well as the leading cause of reduced Quality of Life (QoL) and mortality, with literature indicating that 67% of individuals with a spinal cord injury present with respiratory complications in the acute stage.

The most common respiratory complications are: 1) atelectasis; 2) pneumonia; and 3) respiratory failure. A retrospective review of the patients with acute traumatic spinal cord injuries at C5-T5 level showed a higher prevalence of respiratory complications during the initial hospitalisation just after the injury and suggests the presence of previous respiratory disease, complete motor impairment

(AISA A-B) and coexistent thoracic trauma are a predictor of respiratory complications. Individuals with cervical and higher thoracic spinal cord injuries are more likely to develop respiratory complications, primarily due to diaphragm impairment.

Due to the above, patients have increased rates of infection, poor sputum clearance and inadequate humidification. These complications lead to prolonged admissions, admission to intensive care and considerable healthcare related costs. As such it is essential to develop new management protocols to reduce the occurrence of pulmonary complications

AIRVOTM (a form of non-invasive high flow oxygen therapy, HFOT), which delivers high flow heated and humidified oxygen and air via nasal cannula at a prescribed fraction of inspired oxygen and a maximum flow of 60 L/min, is an attractive alternative to conventional oxygen therapy. Previous studies have shown that HFOT therapy generates a flow-dependent positive airway pressure and improves oxygenation by increasing end-expiratory lung volume, thus suggesting a possible alveolar recruitment associated with high-flow therapy. Although widely used in other clinical areas across the NHS, HFOT delivered via the AIRVOTM system has yet to be evaluated in the spinal cord injury population.

Furthermore, HFNC oxygen therapy has been shown to improved swallowing function in a patient with dysphagia associated with respiratory-muscle paralysis following a SCI, further reducing the risk of aspiration and subsequent infection. It has been hypothesised that the use of HFNC prolongs the patient's apnoea tolerance time during swallowing and hence improves the timing of swallowing.

This study aims to explore the feasibility of using HFOT (delivered via AIRVOTM) therapy and compare to current treatment (conventional oxygen and humidification administration) for patients who have a spinal cord injury. The secondary outcomes will explore any provisional impacts on length of stay, requirement of admission to intensive care, antibiotic use, and physiotherapy requirements including use of cough augmentation e.g., Mechanical Insufflation - Exsufflation.

The results of this proof-of-concept study will be used to further develop local protocols and develop a multi-site research protocol for grant application.

ELIGIBILITY:
Inclusion Criteria:

1. Spinal cord injury between C4 and T4 (Include ASIA A-D)
2. Admitted to spinal injury ward within 24-48hours of injury

Exclusion Criteria:

1. Aged under 18 years
2. 3 or more rib fractures or flail
3. Sternal fracture
4. Concomitant lung injury
5. Unable to gain informed consent from participant
6. Contra-indication to using high flow therapy e.g., undrained pneumothorax, facial fractures, nasal obstruction, CSF leak, suspected or confirmed base of skull fracture, active epistaxis or recent functional endoscopic sinus surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Recruitment rates | 10 days
  This will explore the ability to recruit eligible participants in a timely fashion as per the protocol. It will also capture the participant retainment rates during the study E.g., number of patients recruited, and % of those recruited completing study

SECONDARY OUTCOMES:
To determine the acceptability of the intervention | 10 days
  To see if the protocol can be followed and patients can receive the intervention - do all patients receive the intervention as planned, or is there any cross-over of interventions. E.g. % of participants completing the intervention as planned
Physiotherapy time | 10 days
  Duration (minutes) of physiotherapy intervention during the study period
Frequency of physiotherapy interventions | 10 days
  To understand whether the chosen outcome measures are appropriate - is it appropriate and possible to capture the frequency of physiotherapy intervention during the study period
Pulmonary complications | 10 days
  Incidence of pulmonary complications following spinal cord injury using the brooks-braun classification
Incidence of ICU admission | 10 days
  Incidence of ICU admission during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Paul Twose, Principal Investigator — Cardiff and Vale University Health Board
Locations (1):
- Cardiff and Vale University Health Board, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to for IPD sharing